CLINICAL TRIAL: NCT04308837
Title: A Phase II Trial of Neoadjuvant Laparoscopic Hyperthermic Intraperitoneal Chemotherapy (HIPEC) With Chemoradiation (Carboplatin and Taxol) as First Line Treatment for Patients With Local Regional Advanced Gastric Cancer
Brief Title: A Phase II Trial of Neoadjuvant Laparoscopic Hyperthermic Intraperitoneal Chemotherapy (HIPEC) With Chemoradiation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Spiros Hiotis, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-1101
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Stomach Cancer
Keywords: Phase II Trial; HIPEC; Chemoradiation
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Carboplatin; Dexamethasone; Diphenhydramine; Famotidine; Palonosetron; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: The study design involves a single arm of patients that will all receive the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients With Local Regional Advanced Gastric Cancer (Experimental): Patients with local regional advanced gastric cancer after at least 4 weeks post diagnostic laparoscopy and HIPEC, will receive all of the treatments described in the study protocol.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Famotidine; Drug: Palonosetron; Radiation: 3D conformal or intensity modulated radiotherapy; Procedure: Surgical resection; Radiation: Adjuvant Chemotherapy

INTERVENTIONS:
Drug: Paclitaxel — 50 mg/m2 given by intravenous infusion on days 1, 8, 15, 22 and 29.
Drug: Carboplatin — Carboplatin AUC = 2 given by intravenous infusion on days 1, 8, 15, 22 and 29.
Drug: Dexamethasone — All patients receiving Paclitaxel will receive institutional standard premedications, which include Dexamethasone (10 mg IVPB)
Drug: Diphenhydramine — All patients receiving Paclitaxel will receive institutional standard premedications, which include diphenhydramine (50mg IVP)
Drug: Famotidine — All patients receiving Paclitaxel will receive institutional standard premedications, which include Famotidine (20mg IVPB)
Drug: Palonosetron — All patients receiving Paclitaxel will receive institutional standard premedications, which include Palonosetron (0.25mg IVP)
Radiation: 3D conformal or intensity modulated radiotherapy — Treatment will be given 5 days per week. Photon beams >6 MV are required. Treatment may be delivered either by a 3D conformal technique or IMRT. IMRT via dynamically moving MLCs, step-and-shoot with a multileaf collimator, Rapid Arc, binary multileaf collimator, and tomotherapy are allowed. Proton therapy is not allowed.
  Other Names: IMRT
Procedure: Surgical resection — Surgical resection will constitute subtotal or total gastrectomy (depending on tumor size and location) and D2 lymphadenectomy.
Radiation: Adjuvant Chemotherapy — The patient will begin adjuvant chemotherapy 4-12 weeks after surgery. The adjuvant chemotherapy will consist of FOLFOX every 2 weeks for 6 cycles (i.e. 3 months)

SUMMARY:
Stomach cancer is the fifth most common digestive cancer and third main cause of death from cancer in the world. Modern management of Gastric cancer involves a multi-disciplinary approach involving surgical oncologists, medical oncologists, gastroenterologists and oncological radiologists. The most common clinical approach to Gastric adenocarcinoma is to begin with staging, which usually involves CT scan/ MRI combined with endoscopic US for more accurate T, N staging. Once the patient is deemed to have locally advanced gastric cancer (T3/T4,N0/+), a staging laparoscopy is recommended to rule out obvious or microscopic peritoneal metastatic disease. Additionally, neoadjuvant chemotherapy is initiated and followed by surgery +/- adjuvant radiation and chemotherapy.This protocol involves the addition of neoadjuvant HIPEC at the time of diagnostic laparoscopy as well as neoadjuvant radiation therapy for improved local and systemic control. The goal of this phase II clinical trial is to evaluate the efficacy of a multi-modality approach to treating patients with locally advanced Gastric cancer by incorporating diagnostic laparoscopy with HIPEC, neo-adjuvant chemo-radiotherapy, followed by surgical resection and adjuvant chemotherapy. The trial aims to assess this multi-modality approach in inducing pathological complete response; decreased rates of disease progression during neoadjuvant therapy; and increased overall, disease-free, and peritoneal disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer post endoscopic ultrasound (EUS), staging must be T3/T4
* N0/+, M0. EUS must have been done within 8 weeks of the protocol start.
* Patient must plan to undergo surgical treatment.
* ECOG Scale of Performance Status of 0-2
* Adequate organ and marrow function (leukocytes ≥ 3000/mcl, absolute neutrophil count ≥ 1500, platelets ≥ 100,000/mcl, total bilirubin ≥ 1.5mg/dl (Gilbert's syndrome, then <3.0), AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal, creatinine within normal institutional limits)
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects who have any previous treatment for their cancer.
* Patients with known metastatic disease; this includes patients with clinically apparent or suspected metastasis to sites other than lymph nodes or peritoneal surfaces.
* Subjects with early stage gastric cancer (Stage T1/T2 N0)
* History of allergic reactions attributed to compounds of similar chemical or biological composition to any of the agents being used in this study, including but not limited to: Carboplatin, Taxol, 5-FU, Leucovorin, Mitomycin C.
* Subjects who have received prior radiation to any portion of the abdominal cavity or pelvis are excluded.
* Subjects who have had prior malignancies, except for cured non-melanoma skin cancer, or curatively treated in situ carcinoma of the cervix, or adequately treated malignancies for which there has been no evidence of activity for more than three years.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Subjects with a condition that may interfere with the subjects' ability to understand the requirements of the study.
* Known HIV, Hepatitis B, or Hepatitis C positive patients.
* Patients with active coronary artery disease (defined as unstable angina or a positive cardiac stress test) will be excluded. Subjects with a history of coronary artery disease may be included if they have had a normal stress test within 30 days of enrollment.
* Patients with restrictive or obstructive pulmonary disease that would limit study compliance or place the patient at unacceptable risk for participation in the study will be excluded.
* Patients with a history of cerebrovascular disease that would limit study compliance or place the patient at unacceptable risk for participation in the study will be excluded.
* Subjects with other concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study, or places them at an unacceptable risk for participation in the study, will also be excluded.
* Evidence of extensive intraperitoneal adhesions at the time of surgery which prohibits intraperitoneal therapy, as determined by the operating surgeon.
* Patients with any condition that would precluded the ability to deliver appropriate IP therapy.
* Patients with a life expectancy of less than 12 weeks will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Pathological Response | at time of surgical resection
  The pathological complete response (the lack of all signs of cancer in tissue samples), at the time of surgical resection. This will be determined using a four-category tumor regression score system that evaluates the response of the cancer cells to the treatment. RECIST - Complete Response (CR), Partial Response (PR) Progressive Disease (PD), and Stable Disease (SD)

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 years
  OS is defined as the time from the first dose of study treatment to the date of death (whatever the cause).
Disease-free Survival | 6 years
  The length of time after treatment ends that the patient survives without any signs or symptoms.
Peritoneal Disease-free Survival | 6 years
  The length of time after treatment ends that the patient survives without any peritoneal signs or symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Spiros Hiotis, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai West, New York, New York
  - Mount Sinai St. Luke's, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No